CLINICAL TRIAL: NCT03943121
Title: The Effects of Steroid-eluting Stent Implant for the Treatment of Patients Undergoing Sinus Surgery for Eosinophilic Chronic Rhinosinusitis With Nasal Polyps
Brief Title: The Effects of Steroid-eluting Stent Implant for the Treatment of Eosinophilic Chronic Rhinosinusitis With Nasal Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); China-Japan Union Hospital, Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TR-Stent implant for CRSwNP
Record Dates: First submitted 2019-05-04; First posted 2019-05-09 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-01

CONDITIONS: Patients; Sinusitis; Nasal Polyps
Keywords: Endoscopic sinus surgery; Eosinophilic sinusitis with nasal polyps; Steroid-eluting stent; Randomized Trial
MeSH Terms: conditions — Sinusitis; Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steroid-eluting stent implant (Experimental): The ESS procedure had to be successfully completed without complication on both sides. Steroid-eluting stent were implanted in one side of ethmoid sinus and frontal sinus randomly.
  Interventions: Procedure: Steroid-eluting stent implant
- Without Steroid-eluting stent implant (Sham Comparator): The ESS procedure had to be successfully completed without complication on both sides. The side without the stent is defined as the control side.
  Interventions: Procedure: Without Steroid-eluting stent implant

INTERVENTIONS:
Procedure: Steroid-eluting stent implant — After endoscopic bilateral sinus surgery, the Steroid-eluting stents were randomly implanted in one side of the sinus.
  Arms: Steroid-eluting stent implant
Procedure: Without Steroid-eluting stent implant — After endoscopic bilateral sinus surgery, the Steroid-eluting stents were randomly implanted in one side of the sinus. And the side without the stent is defined as the control side.
  Arms: Without Steroid-eluting stent implant

SUMMARY:
The treatment of eosinophilic sinusitis with nasal polyps is difficult and challenging. After endoscopic sinus surgery(ESS), complications such as edema, scar formation, adhesions, sinus stenosis and recurrence of polyps are prone to occur. Investigators aim to assess the efficacy and safety of Steroid-eluting stent when implanted in sinus in patients following ESS with eosinophilic sinusitis and nasal polyps.The randomized, double-blind, controlled clinical trial enrolled patients with eosinophilic sinusitis and nasal polyps. After endoscopic bilateral sinus surgery, the Steroid-eluting stents were randomly implanted in one side of the sinus and the other side as a control.

Primary outcomes are change in the Lund-Kennedy endoscopic score.The primary outcomes will be measured in baseline, week4,week 8 and week 12. Secondary outcomes include the changes in symptoms measured by Visual analog score and nasal patency (nasal airway resistance and nasal cavity volume), exhaled nasal nitric oxide. The investigators also evaluate change in inflammatory cytokines (interleukin(IL)-4, IL-5, IL-8, IL-17, IL-22, IL-25, interferon-γ, tumor necrosis factor-α, transforming growth factor-β, Leukotriene,Eotaxin) in nasal secretions. The secondary outcomes will be measured in baseline, week4, week8 and week12. Mucosal pathology assessment will be performed at 4 weeks postoperatively.Sinus CT scan will be conducted at 8 weeks after surgery. Changes in serum cortisol are monitored at baseline,week4 and week12 postoperatively. All adverse events are recorded throughout the experiment

ELIGIBILITY:
Inclusion Criteria:

1. Subjects were 18-65 years old, male or non-pregnant women;
2. Understands the purpose and procedures of the trial and voluntarily signs the informed consent form;
3. Subjects must meet the guidelines for the diagnosis of chronic sinusitis and nasal polyps (EPOS2012), diagnosed with bilateral chronic sinusitis and nasal polyps. Histopathological examination showed a percentage of eosinophils >27%.
4. Planned sinus surgery includes bilateral sinus opening surgery, the same equipment should be used on both sides, FESS surgery must be successfully completed, and no complications;
5. Female subjects were not in the lactation period during the screening visit and had no breastfeeding and pregnancy plan for up to 1 year after the start of the operation;
6. Subjects did not participate in other clinical trials for the first three months and agreed not to participate in other clinical trials until the end of the trial was reached.

Exclusion Criteria:

1. The subject has a known allergic reaction or contraindication to the device material and its degradation products (mamethasone citrate, L-polylactic acid, racemic polylactic acid, lactide lactate, lactic acid);
2. Subjects need long-term oral steroid drugs;
3. The subject is receiving immunotherapy for immunosuppressive or autoimmune diseases;
4. Subjects have severe diabetes or Hypertension;
5. Subjects have suffered or are suffering from glaucoma or ocular hypertension;
6. Subjects have cataracts;
7. Patients with acute bacterial sinusitis and acute fungal sinusitis;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
The change in the Lund-Kennedy endoscopic score | Baseline, week4,week 8 and week 12
  We used the Lund-Kennedy endoscopic scoring system to measure the patient's nasal cavity based on fi there were edema, vesicles, adhesions, scars and polyps.

SECONDARY OUTCOMES:
The changes in nasal symptoms | Baseline, week2, week4, week8, week12
  Nasal symptoms measured by Visual analog score. The four nasal symptoms (nasal obstruction, rhinorrhea, headache and olfactory disorder) involved in assigning the total nasal symptom score(TNSS). The symptoms are graded on a10-point scale (0 = no symptoms;10 = most severe symptoms).
Nasal patency | Baseline, week4, week8 and week12
  Acoustic rhinometry was performed to measure the total nasal cavity volume (cm³) and Rhinomanometer was used to measure the total nasal airway resistance (Pa·cm-³·s-1) .
Exhaled nasal nitric oxide | Baseline, week4, week8 and week12
  Measure exhaled nasal nitric oxide (nNO). Briefly, NO-free air was aspirated through the nasal cavity at a flow rate of 50 ml/s. The subject exhaled against the air-resistance, resulting in an intraoral pressure to close the velum and prevent mixture of oral and nasal gas. Nasal gas from this circuit was continuously routed in part directly into the analyser for determination of nNO, and the level of nNO(ppb) was calculated from a plateau lasting for at least 3s.

OTHER OUTCOMES:
Inflammatory cytokines (interleukin(IL)-4, IL-5, IL-8, IL-17, IL-22, IL-25, interferon-γ, tumor necrosis factor-α, transforming growth factor-β, Leukotriene,Eotaxin) in nasal secretions. | Baseline, week4, week8 and week12
  The change of inflammatory cytokines (interleukin(IL)-4, IL-5, IL-8, IL-17, IL-22, IL-25, interferon-γ, tumor necrosis factor-α, transforming growth factor(TGF)-β1, TGF-β2, TGF-β3,Chemokine, Eotaxin) in nasal secretions as secondary outcomes. Nasal secretions were obtained by inserting a postoperative sinus pack in the nasal cavity (acupuncture side) for five minutes. The quantity of secretions was determined by comparing the weight of the sponges before and after insertion and 2 ml of 0.9% sodium chloride solution was added to each sponge. The sponges were stored at 4°C for two hours and the nasal secretions were recovered from the sponges by centrifugation at 1500 g for 15 minutes at 4°C. The supernatants were separated and stored in aliquots at -20°C until further analysis. The levels of inflammatory cytokines (pg/g) were analysed using the Luminex System.
Mucosal pathology assessment | Week4
  We obtained nasal mucosa and performed pathological observations to observe changes in the level of inflammatory and changes in the number and quantity of inflammatory cells.
Sinus CT scan | Week 8
  Using CT scanning, we observed changes in the Lund-Mackey scores of bilateral nasal sinuses .
Changes in serum cortisol | Baseline,week4 and week12
  We validate the safety of stent implantation by examining serum cortisol.
Adverse events | Week2, week4, week8, week12
  During the progress of the experiment, we pay attention to the findings of patients with or without severe reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China